CLINICAL TRIAL: NCT03829956
Title: The Efficacy of Intra-oral Neuromuscular Stimulation Training on Primary Snoring
Brief Title: Intraoral Tongue Stimulation for Treatment of Primary Snoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Signifier Medical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Snoozeal
Record Dates: First submitted 2017-01-13; First posted 2019-02-04 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Snoring; Obstructive Sleep Apnea
Keywords: snoring; obstructive sleep apnoea; hypopnoea
MeSH Terms: conditions — Snoring; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Snoring and mild OSA (Other): This cohort of participants has been diagnosed with primary snoring or mild obstruction sleep apnoea. A medical device (intra-oral tongue stimulation device) will be introduced for 6 weeks and the effects will be assessed by comparing the outcome measures before and after the intervention.
  Interventions: Device: Intraoral tongue stimulator (Snoozeal)

INTERVENTIONS:
Device: Intraoral tongue stimulator (Snoozeal) — Electrical stimulation of the tongue muscle to improve muscle tone to treat primary snoring and mild obstructive sleep apnea.

SUMMARY:
Intraoral Neuromuscular Training for Treatment of Snoring

Objective

Studies show that improving pharyngeal muscle tone can ameliorate obstructive sleep apnoea (OSA) and snoring. The study uses an intra-oral stimulation device (SnooZeal) aimed at a population of snorers. The aim of this study is to assess the efficacy of intra-oral neuromuscular stimulation training during wakefulness on snoring.

Methods

This is a prospective study, recruiting up to 200 patients from the sleep clinics.

In this study, subjects will use the intra-oral stimulation device once a day for 20 minutes each time for a period of 6 weeks. During these 6 weeks, subjects will complete a daily diary of the device use and any side effects or adverse events. Partners also complete a daily snoring score.

Subjects will be followed-up for a further 2 weeks after treatment. They will complete Pittsburgh Sleep Quality Index (PSQI) and subjective sleep quality questionnaires for a further 2 weeks. Partners will also complete the post treatment snoring scores. Sleep study will be repeated.

Outcome measures

The objective evaluation will be based on pre- and post-treatment sleep studies, visual analogue scale (VAS) snoring scores, PSQI and subjective sleep quality questionnaire. All side effects and adverse events will be reported and acted upon according to the risk management structure.

DETAILED DESCRIPTION:
Aim/ Objective

The aim of this study will be to assess the efficacy of transoral neuromuscular stimulation training during wakefulness on snoring.

Patients and Methods

This is a prospective observational study, recruiting patients from the sleep clinics at the Department of Otorhinolaryngology, Head and Neck Surgery in Queen's Hospital, Barking, Havering and Redbridge University Hospitals National Health Service (NHS) Trust

Sample size planned is up to 200 participants.

Study Protocol

A. Screening Participants will be identified from Queen's Hospital, Barking, Havering and Redbridge NHS Trust. There will be a screening phone call to ensure suitability based on an inclusion criterion and offer first line information about the trial. If suitable, participants will be given a written information sheet and invited to undertake a 2 day home sleep study (using WatchPAT). If the average apnea-hypopnea index (AHI) from these 2 days is below 15/h, the participants will be invited for a clinical examination.

B. Recruitment visit

* Clinical airway examination by Ear, Nose and Throat (ENT) consultant
* Review of inclusion and exclusion criteria
* Informed consent
* Inclusion into trial

C. Pre-therapy period (day -14 to -1):

* Bed partner daily subjective assessment of snoring (Visual Analogue Scale - participant's bed partner will be required to complete daily visual analogue scoring of the participant's snoring, with 1 being "no snoring" and 10 being "intolerable snoring")
* Oral examination (detailed examination by dentist to document pre-therapy oral state
* Participant and bed partner to complete sleep quality questionnaires (Pittsburgh Sleep Quality Index, Epsworth sleepiness score (ESS) and subjective sleep quality questionnaire) on Day -1

D. Therapy phase (day 1-42)

* Face-to-face meeting, instruction on use of the intraoral device
* Participant to use the Snoozeal device for 20 minutes once daily
* Bed partner daily subjective assessment of snoring (VAS)
* Participant daily assessment of side effects/adverse events and time of use
* Participant and bed partner to complete Sleep quality Questionnaires (Pittsburgh Sleep Quality Index, Epsworth sleepiness score and subjective sleep quality questionnaire) at day 42
* Weekly follow up phone call from research team to confirm compliance. Compliance will also be cross checked using the total time of use recorded by the device.

E. End of Therapy Review (day 43 - 49)

* Review of device integrity by visual inspection
* Oral examination (detailed examination by dentist to document post therapy oral state)
* Repeat Sleep Study - 2 night sleep study with WatchPAT

F. Follow Up phase (day 43-56)

* Participant advised to stop using device
* Bed partner daily subjective assessment of snoring (VAS)
* Subject and bed partner to complete Sleep quality Questionnaires (Pittsburgh Sleep Quality Index, Epworth sleepiness score and subjective sleep quality questionnaire) at day 56

G. Post Therapy Review (day 57)

* Face-to-face meeting and feedback
* Collection of participant data sheets
* Participant subjective overall assessment

Data Analysis

The pre and post sleep studies will be performed using WatchPAT. Parameters recorded: saturation, AHI, snoring sound parameters.

AHI will be identified and analyzed by WatchPAT data and software. The WatchPat is an approved FDA sleep study device. Snoring will be quantified subjectively by both the bed partner using a visual analog score, and objectively during the home sleep study as frequency of snores (number of snores / hours of sleep) and % total sleep time spent snoring. Sleep quality will be quantified subjectively by PSQI score. Sleepiness will be quantified subjectively by ESS score.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above at entry into study
* Subjects must have a live-in partner
* > 6 months history of habitual snoring (>5 days per week)

Exclusion Criteria:

* Body Mass Index > 35
* Apnoea-Hypopnoea Index >15
* Symptomatic nasal pathology
* Tonsil Hypertrophy (Tonsil size > Grade 2)
* Tongue or lip piercing
* Pacemaker or implanted medical electrical devices
* Previous oral surgery for snoring
* Relevant facial skeletal abnormalities
* Certain oral disease/conditions (see Appendix 3)
* Any criteria that, in the opinion of the investigator, would make the participant unsuitable for the study due to inability to complete required study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

PRIMARY OUTCOMES:
Reduction in snoring levels greater than 40dB | Change between pre-therapy (day -14 to -1) and end of therapy (day 43-49)
  Reduction of 20 % in the percentage of time spent snoring at levels greater than 40 dB. This will be achieved using WatchPat (510K - K161579) sleep studies
Visual analogue scale (VAS) snoring scores | Change between average of pre-therapy (day -14 to day -1), during therapy (day 29 to 42) and post therapy (day 43 to 56)
  Visual analogue scale (VAS) of snoring is a subjective assessment of the participant's severity of scoring by their partner on a scale of 1 - 10 (1 being no snoring, 10 being intolerable snoring). This assessment will be done on a daily basis for the 2 weeks prior to intervention, 6 weeks of intervention and 2 weeks post intervention.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Change between pre-therapy (day -1) and post therapy (day 56)
  Pittsburgh Sleep Quality Index is a self-report questionnaire that is completed by the participants at day -1 (pre-therapy), day 42 (end of therapy) and day 56 (post therapy). The questions are multiple choice questions with the answers based on participants' usual sleep habits during the last four weeks. The outcome is assessed based on the evaluation of the change in responses before and after therapy. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Epworth Sleepiness Scale (ESS) | Change between pre-therapy (day -1) and post therapy (day 56)
  The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The score can range from 0 to 24, with a higher score indicating a higher level of daytime sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Bhik Kotecha, Principal Investigator — University College London Hospitals
Locations (1):
- Redbridge, Barking and Havering NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nokes B, Baptista PM, de Apodaca PMR, Carrasco-Llatas M, Fernandez S, Kotecha B, Wong PY, Zhang H, Hassaan A, Malhotra A. Transoral awake state neuromuscular electrical stimulation therapy for mild obstructive sleep apnea. Sleep Breath. 2023 May;27(2):527-534. doi: 10.1007/s11325-022-02644-9. Epub 2022 May 27. PMID 35624401
- [Derived] Kotecha B, Wong PY, Zhang H, Hassaan A. A novel intraoral neuromuscular stimulation device for treating sleep-disordered breathing. Sleep Breath. 2021 Dec;25(4):2083-2090. doi: 10.1007/s11325-021-02355-7. Epub 2021 Mar 26. PMID 33772397

DOCUMENTS (2):
  • Study Protocol (2018-12-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT03829956/Prot_000.pdf
  • Informed Consent Form (2018-12-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT03829956/ICF_001.pdf